CLINICAL TRIAL: NCT05031520
Title: A Single Center Study of Perivascular Coronary Inflammation in Patients With Myocardial Ischemia or Infarction With Non-Obstructive Coronary Arteries
Brief Title: PericOronary INflammaTion in Non-Obstructive Coronary Artery Disease
Acronym: POINT-NOCAD
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to funding expiration.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-00764
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Non-Obstructive Coronary Atherosclerosis
MeSH Terms: interventions — Iopamidol; Nitroglycerin; Metoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: Participants will be identified by review of the cardiac catheterization laboratory schedule each day by the principal investigator, a co-investigator, or a research coordinator. Participants with no obstructive CAD and completed microvascular testing will undergo a research CCTA.
  Interventions: Procedure: Coronary computed tomography angiography (CCTA); Drug: Isovue; Drug: Nitroglycerin; Drug: Metoprolol

INTERVENTIONS:
Procedure: Coronary computed tomography angiography (CCTA) — Participants will undergo CCTA. CCTA performed in this study will be technically identical to CCTA that is commonly performed in clinical practice, for which safety profiles are well defined. Guidelines implemented by the National Institutes of Health Radiation Exposure Committee will be followed. Major risks of CCTA include exposure to ionizing radiation, the requirement for intravenous catheter placement and contrast media administration, and side effects of beta-blockers and nitrates that may be used for vasodilation and heart rate control to optimize CCTA image quality.
Drug: Isovue — CCTA requires intravenous catheter placement and the administration of iodinated contrast media (Isovue).
Drug: Nitroglycerin — Medication to promote coronary vasodilation during the CCTA may be administered immediately prior to CCTA to optimize image quality
Drug: Metoprolol — Medication to promote heart rate reduction during the CCTA may be administered immediately prior to CCTA to optimize image quality

SUMMARY:
Among patients with ischemic heart disease who are referred for coronary angiography, a substantial proportion have non-obstructive coronary artery disease (CAD). Myocardial infarction (MI) with non-obstructive coronary artery disease (MINOCA) accounts for 5-20% of patients with MI and preferentially affects women. MINOCA pathogenesis is varied and may include atherosclerotic plaque rupture, plaque erosion with thrombosis, vasospasm, embolization, dissection or a combination of mechanisms. Other patients may have clinically unrecognized myocarditis, or takotsubo syndrome masquerading as MI. Among patients referred for coronary angiography for the evaluation of stable ischemic heart disease, non-obstructive CAD is present in up to ~30% of men and ~60% of women. Stable ischemia with non-obstructive coronary arteries (INOCA) may be due to coronary microvascular dysfunction in up to 40% of these patients. Our understanding of mechanisms of MINOCA and INOCA remain incomplete. Coronary inflammation has been hypothesized as a potential mechanism contributing to coronary spasm in MINOCA and microvascular disease in INOCA.

DETAILED DESCRIPTION:
The PericOronary INflammaTion in Non-Obstructive Coronary Artery Disease (POINT-NOCAD) study is a single-center diagnostic, observational study enrolling men and women with MINOCA or INOCA who are planned to undergo (or underwent) clinically indicated coronary angiography. The research plan is to evaluate coronary inflammation, as measured by the perivascular coronary fat attenuation index from non-invasive coronary computed tomography angiography (CCTA), in patients with MINOCA and INOCA.

ELIGIBILITY:
Inclusion Criteria:

* Adult age ≥18 years referred for clinically indicated coronary angiography
* Stable ischemic heart disease OR acute myocardial infarction as the indication for coronary angiography

Exclusion Criteria:

Clinical Exclusion criteria:

* Estimated glomerular filtration rate < 45 mL/min
* History of allergic reaction to iodinated contrast media
* Pregnancy

Angiographic / Post-Cath Exclusion criteria:

* Obstructive CAD (≥50% luminal obstruction in ≥1 major epicardial coronary arteries by invasive coronary angiography)
* Allergic reaction to iodinated contrast media

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the NYU Langone Health Tisch/Kimmel Cardiac Catheterization Laboratory or the Bellevue Cardiac Catheterization laboratory will be screened and approached for consent if the patient's treating provider is amenable to their participation in the research study and if the patient is eligible for enrollment based on the eligibility criteria prior to clinically indicated cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Perivascular coronary fat attenuation will be significantly greater in MINOCA patients compared with INOCA patients | Visit 1, Day 0
  Images obtained from the CCTA will be used to calculate perivascular FAI, measured around the proximal left anterior descending artery and in the right coronary artery, in the proximal 10 to 50 mm of the vessel. For each coronary vessel, will define the weighted mean attenuation of all adipose tissue-containing voxels (-190 to -30 Hounsfield units [HU]) located within a radial distance from the outer vessel wall equal to the diameter of the respective vessel.
Perivascular coronary fat attenuation will be greater in INOCA patients with versus without coronary microvascular disease | Visit 1, Day 0
  Images obtained from the CCTA will be used to calculate perivascular FAI, measured around the proximal left anterior descending artery and in the right coronary artery, in the proximal 10 to 50 mm of the vessel. For each coronary vessel, will define the weighted mean attenuation of all adipose tissue-containing voxels (-190 to -30 Hounsfield units [HU]) located within a radial distance from the outer vessel wall equal to the diameter of the respective vessel.
Perivascular coronary fat attenuation in patients with MINOCA will be greatest in the culprit coronary vessels with evidence of acute plaque disruption. | Visit 1, Day 0
  Images obtained from the CCTA will be used to calculate perivascular FAI, measured around the proximal left anterior descending artery and in the right coronary artery, in the proximal 10 to 50 mm of the vessel. For each coronary vessel, will define the weighted mean attenuation of all adipose tissue-containing voxels (-190 to -30 Hounsfield units [HU]) located within a radial distance from the outer vessel wall equal to the diameter of the respective vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Smilowitz, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Nathaniel.Smilowitz@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05031520/ICF_000.pdf